CLINICAL TRIAL: NCT02099396
Title: A Clinical Trial on Efficacy and Safety for Lobaplatin and Gemcitabine in Combination With Docetaxel in the Second-line Treatments on Advanced Osteosarcoma
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: China Association of Osteosarcoma Chemotherapy (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ChinaAOC-2014-001
Record Dates: First submitted 2014-03-26; First posted 2014-03-28 (Estimated); Last update posted 2014-03-28 (Estimated); Status verified 2014-03

CONDITIONS: Lobaplatin and Gemcitabine in Combination, Second-line Treatments on Advanced Osteosarcoma
Keywords: PFS,efficacy and safety,lobaplatin and gemcitabine in combination, second-line treatments on advanced osteosarcoma

ARMS (2):
- docetaxel+lobaplatin (Experimental): Pretreatment: 15 mg dexamethasone is administered orally every day since one day before administration with docetaxel for continuous three days. Dexamethasone 10 mg i.v. and promethazine 25mg im are administered 30 min before administration with docetaxel to prevent anaphylactic responses.
  Intravenous infusion with docetaxel 75mg/m2 for one hour is carried out on the first day of each cycle for 21 days; intravenous infusion with lobaplatin 30 mg/m2 for two hours is carried out on the second day; q3wkb
  Interventions: Drug: Docetaxel+lobaplatin
- gemcitabine+lobaplatin (Experimental): Pretreatment: 15 mg dexamethasone is administered orally every day since one day before administration with docetaxel for continuous three days. Dexamethasone 10 mg i.v. and promethazine 25mg im are administered 30 min before administration with docetaxel to prevent anaphylactic responses.
  Intravenous infusion with gemcitabine 675mg/m2 for 90 min is carried out on the first day and the eighth day of each cycle for 21 days; intravenous infusion with lobaplatin 30 mg/m2 for two hours is carried out; intravenous infusion with docetaxel 75mg/m2 for one hour is carried out on the first day; q3wkb
  Interventions: Drug: Gemcitabine+lobaplatin

INTERVENTIONS:
Drug: Docetaxel+lobaplatin
  Arms: docetaxel+lobaplatin
Drug: Gemcitabine+lobaplatin
  Arms: gemcitabine+lobaplatin

SUMMARY:
The purpose was to evaluate efficacy, safety and effects on survival for lobaplatin and Gemcitabine in combination with Docetaxel, which can provide a kind of completely new second-line chemotherapy program for osteosarcoma patients in aggressive-phase, provide accurate and reliable evidence-based results for clinical applications of lobaplatin in osteosarcoma patients as one of the third-generation of platinum drugs, and further consummate and enrich clinical practice guidance on osteosarcoma all over the world.

ELIGIBILITY:
Inclusion Criteria:

- 1. 8-40 years old, male or female

2. Osteosarcoma in aggressive-phase confirmed by histopathology. Local tumors and isolated pulmonary foci must be confirmed by pathological diagnosis, and pathological examinations are not required for pulmonary multiple metastatic tumors

(Definition for osteosarcoma in aggressive-phase:

1. Primary tumors or locally recurrent tumors that are impossible to cure or it can be radically cured by amputation but patients refuse
2. osteosarcoma showing distal metastasis, metastatic tumors that are unable for radical cure by operations or other local therapeutic methods (such as stereotaxic radiosurgery, argon-helium knife, ultrasonic focusing knife)
3. patients refuse or could not tolerate operations or other local treatments for both primary tumors and metastatic tumors.)

   But the patients as below are not included:
   1. Pulmonary metastasis complicated with more than three osseous metastasis foci at the same time
   2. Local recurrent foci of bigger than 200mm3
   3. More than three pulmonary metastasis foci of bigger than 3cm
   4. Diffusive pulmonary metastasis
   5. More than 10 metastatic foci of bigger than 1 cm in both lungs
   6. Intracranial metastasis
   7. Multiple metastasis in pelvis
   8. Formation of tumor embolus in great vessels (thigh vessels, iliac vessels, peritoneal cavity vessels, vessels in armpits, infraclavicular vessels)
   9. Coelom effusion 3. Patients fails in the treatments with the first-line chemotherapeutics for osteosarcoma (HD-MTX, ADM, DDP, IFO), those having ever used at least three kinds of first-line drugs.

      4. Patients showing progression of disease within six months after neoadjuvant chemotherapy or adjunctive chemotherapy for osteosarcoma as well as first-line chemotherapy, permission from the subjects or their legal representatives should be obtained for patients showing progression of disease for more than six months.

      5. Measurable foci are detected at baseline according to RECIST 1.1 edition. 6. ECOG physical efficiency score at 0-1, anticipated life span for more than three months.

      7. Recovery from previous treatments: according to NCI-CTC AE 4.0 edition, all of the adverse reactions (except baldness) recover to grade one or even lower.

      8. Peripheral hemogram and blood biochemical indicators as follows indicate proper organ functions: Hemoglobin (Hb)≥ 90g/L, Neutrophilic granulocyte (ANC)≥1.5×109/L, Blood platelet count (Plt)≥ 80×109/L, Serum creatinine (Cr)≤ 1.5×upper normal limit (ULN), blood urea nitrogen (BUN)≤ 2.5×upper normal limit (ULN); Total bilirubin (TB)≤ ULN; Alkaline phosphatase (ALP)≤ 2.5×ULN; Aspartate aminotransferase (AST) and glutamate pyruvate transaminase (ALT)≤ 2.5×ULN; albumen (ALB)≥ 25 g/L。 9. Pregnancy test (urinary β-HCG) negative (suitable for women in reproductive life having sexual activities).

      10. Informed consent (or signed by their legal representatives) are signed to testify that they understand the purpose of the study and the operations required in the study, and they are willing to participate in the present study, and the subjects below 18 year old should sign the informed consent for minors.

      Exclusion Criteria:
      * 1. Previous exposure to lobaplatin / docetaxel, lobaplatin / gemcitabine, docetaxel / gemcitabine.

        2. Within three weeks after the last systemic cytotoxic drug medication, radiotherapy or treatments with any test drug.

        3. Suffering from other malignant tumors during the past three years. Exceptions: skin basal cell carcinoma or nonmetastatic squamous cell carcinoma, carcinoma in situ of uterine cervix, or FIGO period 1 cervical cancer.

        4. Previously known metastasis to central nervous system. 5. Myocardial infarction within six months before inclusion, grade II or higher cardiac failure defined in New York Cardiac Association, uncontrolled angina pectoris, uncontrolled severe ventricular arrhythmia, pericardial diseases with clinical significance, or electrocardiogram indicates acute ischemia or abnormalities in reactive conducting system.

        6. Uncontrolled complications, including but not confined to: poorly controlled hypertension or diabetes, persistent reactive infections, or psychological diseases or social situations that may affect the compliance of the subjects to the research.

        7. Previously known allergic reactions, hypersensitivity or intolerance to lobaplatin, docetaxel, gemcitabine or adjuvant.

        8. Women in pregnancy or lactation. 9. Any situation pointed by the researcher that may impair the subjects or lead to incapability to meet with or implement the requirements of the research.

Ages: 8 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 100 (Estimated)
Dates: Start 2014-04; Primary Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
progression free survival (PFS) | 2 years
  Major parameter: progression free survival (PFS) Progression free survival (PFS): it refers to the period from the day of randomization in the groups to any progression of disease or death with records.

SECONDARY OUTCOMES:
Minor parameters: objective remission rate (ORR) | 2 years
  Overall survival (OS): it refers to the period from the date of randomization in the groups to death induced by any reason with records. The ending date of last correspondence should be recorded for all of the subjects lost from follow-ups before termination of the clinical trials or quit from the tests. The last date for survival will be recorded as the ending for the subjects still accepting treatments.
Minor parameters: overall survival (OS), safety. | 2 years
  Objective remission rate (ORR): it refers to the percentage of patients for whom tumors decrease to certain sizes and maintain for a period, including CR and PR cases. The criteria for evaluations on therapeutic efficacy are divided into complete remission (CR), partial remission (PR), stable disease (SD) and progression of disease (PD) according to the RECIST criteria (please refer to attachment 1 for details).